CLINICAL TRIAL: NCT02375217
Title: "Low Dose Sugammadex Combined With Neostigmine and Glycopyrrolate Versus Full Dose Sugammadex for Reversal of Rocuronium-induced Neuromuscular Blockade: a Cost Saving Strategy"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Marie Awad, Professor of clinical Specialty, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANES.MA.14
Record Dates: First submitted 2015-02-11; First posted 2015-03-02 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Anesthesia Recovery
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 : (NS) (Active Comparator): Group 1 Drug combination:
  patients receive half of the recommended dose of sugammadex plus dose of neostigmine"
  1. Sugammadex IV= -1 mg/kg( moderate NMB) or
     * 2 mg/kg (deep NMB)
  2. neostigmine IV = 50mcg/kg
  3. glycopyrrolate 10 mcg/kg
  Interventions: Drug: Sugammadex; Drug: Neostigmine; Drug: glycopyrrolate
- Group 2 : (S) (Active Comparator): patients receive Full recommended dose of sugammadex
  Sugammadex IV= 2mg/kg (Moderate NMB) 4mg/kg ( Deep NMB)
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — half dose
  Arms: Group 1 : (NS)
Drug: Sugammadex — full dose
  Arms: Group 2 : (S)
Drug: Neostigmine — IV = 50mcg/kg
  Arms: Group 1 : (NS)
Drug: glycopyrrolate
  Arms: Group 1 : (NS)

SUMMARY:
Prospective Randomized non inferiority Trial involving adult patients undergoing elective surgery under general anesthesia.56 Patients will be enrolled in 2 groups : full dose sugammadex vs half dose sugammadex for reversal of NMB.

DETAILED DESCRIPTION:
The investigators' aim is to prove that half dose sugammadex in combination with neostigmine 0.05 mg/kg is non-inferior to the recommended dose of sugammadex for the reversal of deep ( absence of Trian of Four response :TOF) or moderate ( TOF 1 or 2 twiches) muscle paralysis in patients undergoing surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70
* ASA class I, II, and III
* undergoing surgery under balanced general anesthesia requiring the use of muscle relaxants throughout the surgery

Exclusion Criteria:

* patients undergoing emergency surgeries
* pregnant patients
* patients with end stage renal disease or chronic kidney disease(GFR less than 60)
* patients with allergy to sugammadex or who had previous complications or side effects from previous sugammadex administration
* patients' refusal
* patients with allergy to recuronium

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
TOF ratio of 0.9 | within 5 minutes

SECONDARY OUTCOMES:
the time to return of TOF ratio to 0.9 and the time till extubation | within 10 minutes
Residual neuro-muscular blockade | within 10 to 180 mins
  Post Anesthesia recovery unit

CONTACTS AND LOCATIONS:
Overall Officials: Marie Mn Aouad,, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- AUBMC, Beirut, Lebanon

REFERENCES:
- [Derived] Aouad MT, Alfahel WS, Kaddoum RN, Siddik-Sayyid SM. Half dose sugammadex combined with neostigmine is non-inferior to full dose sugammadex for reversal of rocuronium-induced deep neuromuscular blockade: a cost-saving strategy. BMC Anesthesiol. 2017 Apr 11;17(1):57. doi: 10.1186/s12871-017-0348-9. PMID 28399799